CLINICAL TRIAL: NCT03921476
Title: Acne and Mood: Impact of Treatment on Depression, Anxiety, and Sexual Function
Status: Withdrawn | Type: Observational
Why Stopped: Investigator left Northwestern University
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Stephanie Rangel, Research Assistant Professor of Dermatology, Northwestern University
Other Study IDs: BJS07172018
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects on spironolactone for a diagnosis of acne vulgaris: Female subjects between 18 and 65 years of age currently taking spironolactone for a diagnosis of acne vulgaris
  Interventions: Other: Online survey
- Subjects on oral antibiotics for a diagnosis of acne vulgaris: Female subjects between 18 and 65 years of age currently taking oral antibiotics for a diagnosis of acne vulgaris
  Interventions: Other: Online survey

INTERVENTIONS:
Other: Online survey — Online survey completion through Northwestern's REDCap

SUMMARY:
This study seeks to examine if there is any relationship between spironolactone use prescribed for acne vulgaris and depression, anxiety, and/or sexual function.

ELIGIBILITY:
Inclusion Criteria:

Female subjects between 18 and 65 years of age currently taking spironolactone for a diagnosis of acne vulgaris

OR

Female subjects between 18 and 65 years of age currently taking oral antibiotics for a diagnosis of acne vulgaris

AND Subjects able to complete an online survey in English

Exclusion Criteria:

Subjects less than 18 years of age or older than 65 years of age Subjects that have ever been diagnosed with any mood disorder by a clinician prior to starting spironolactone (history of mood disorder or current mood disorder) Subjects taking hormonal contraception (including but not limited to oral contraceptive pills) for a duration of less than 6 months Subjects that have ever been diagnosed with any type of sexual dysfunction prior to starting spironolactone Subjects not able to complete an online survey in English Subjects taking oral isotretinoin for a diagnosis of acne Subjects that are currently pregnant

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Biologically female subjects
Study Population: Female patients who have acne vulgaris being treated with spironolactone or oral antibiotics.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent correlation between spironolactone use for acne vulgaris and increased prevalence of depression. | one week
  Score for depression from subject reported Dermatology Life Quality Index (DLQI) survey
Percent correlation between spironolactone use for acne vulgaris and increased prevalence of anxiety. | two weeks
  Score for depression from subject reported Generalized Anxiety Disorder (GAD-7) survey
Percent correlation between spironolactone use for acne vulgaris and increased prevalence of sexual dysfunction. | four weeks
  Score for depression from subject reported Female Sexual Function Index (FSFI) survey.

CONTACTS AND LOCATIONS:
Overall Officials: Bethanee Schlosser, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No